CLINICAL TRIAL: NCT06022991
Title: TARGET Study: faThers And paRtners in Family inteGrated carE sTudy- A Prospective Multicentre Multiphase Study Investigating Father/Partner Involvement in Family Integrated Care in Neonatal Units
Brief Title: Fathers and Partners in Family Integrated Care Study
Acronym: TARGET
Status: Recruiting | Type: Observational
Sponsor: Homerton University Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 152449
Record Dates: First submitted 2022-07-27; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Mental Health Wellness 1; Premature Birth
Keywords: Father/partner wellbeing; Maternal wellbeing; Paternal infant engagement; NICU; Family integrated care (FICare)
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
AIMS: The primary aim is to investigate the impact of enhancing father/partner engagement in FICare of preterm infants on their mental health (MH) up to 6 weeks post discharge. Secondary aims are to investigate the impact on maternal MH.

METHOD and ANALYSIS: This is a two-phase study: Phase-1 to gather baseline information and Phase-2 to assess the impact of improved father/partner engagement in FICare involving two NUs (a tertiary and level 2). 20 families of infants born at <33 weeks will be studied in each phase (40 fathers, 40 mothers, 40 babies).

Father/partner MH will be assessed using validated questionnaires: Generalised Anxiety Disorder Assessment (GAD-7), Patient Health Questionnaire (PHQ-9), Parental Stressor Scale: NICU (PSS:NICU), and by semi-structured qualitative interviews. Similarly, mothers will be assessed by the same questionnaires and focus groups.

The Neonatal DadPad materials will be updated using information from phase 1 study, systematic review of Fathers experiences of FICare and advice from parent advisory group. Father's engagement in FICare will be enhanced using Neonatal DadPad information booklet and app, father-specific peer support and bitesize teaching on caring for NU babies (Phase 2).

Thematic analysis of the qualitative data will be performed. Phase 1 and Phase 2 study findings will be compared by performing appropriate statistical analysis.

DETAILED DESCRIPTION:
BACKGROUND: Family-integrated care (FIC) is a culture whereby parents are viewed as collaborators in their baby's care in neonatal units. This can be challenging for fathers/non-birthing partners as they face competing demands on their time to try and allow the mother to focus on her baby.

KEY AIMS AND OBJECTIVES:

Aims To undertake an in-depth longitudinal study of the engagement of fathers/partners in FiCare and their experience and mental health (MH) from neonatal unit admission to 6 weeks post discharge of their premature baby born at <33 weeks gestation.

Objectives:

1. To assess baseline fathers' experiences in the NU, their involvement in FICare, and MH status during babies NU admission up to 6 weeks post-discharge
2. To conduct systematic review (SR) of published articles on 'Fathers and FiCare in NU' and 'Fathers' MH in the NU'.
3. To develop a programme to enhance involvement of fathers in FiCare.
4. To introduce the programme developed to enhance fathers' involvement in FiCare and explore their experiences and effect on their MH.

Methods

Study design:

This is a prospective multi-centre and multi-phase pilot study. Phase 1 will assess baseline fathers' experiences in the NU, their involvement in FICare and MH status during babies' NU admission up to 6 weeks post-discharge. Simultaneously, a systematic review of fathers' involvement in FICare and their MH outcomes will be conducted. A programme to enhance the involvement of fathers in FICare will be developed using information from phase-1 study, systematic review, existing DadPad app and advice from parent advisory group (PAG). In phase-2 study, enhanced father involvement programme in FICare will be implemented and similar assessments as in phase-1 will be conducted (Figure 1). Regular debrief sessions, and research updates/newsletters to keep staff engaged and supportive of the project will be provided. This support will be continued throughout the study.

Study Centres: The study will be conducted at a tertiary neonatal unit (level 3) and a local neonatal unit (level 2) as defined by the Department of Health, from East London, UK. The Parent Advisory Group (PAG) will help to update the existing Neonatal DadPad app and booklet. They will provide support in finalising topic guides for fathers' education classes for phase-2 study. The PAG will also support in dissemination of the study findings to research participants and the wider neonatal community.

Phase 1 study. Baseline Data Collection: 9 months

1. Prior to the introduction of the study to wider NU clinical staff members, staff knowledge, experiences and opinions about the role of fathers and FICare will be assessed by a questionnaire.
2. Once a parent is recruited, the Parental Stressor Scale: NICU (PSS:NICU)20, and MH questionnaires (Generalised Anxiety Disorder Assessment (GAD-7)21 and, Patient Health Questionnaire (PHQ-922)) will be given to complete within 7 days.
3. Fathers/partners will be invited to participate in 2 semi-structured interviews, within 2 weeks of recruitment and immediately prior to discharge. The interviews will explore their MH, experiences of bonding with baby, understanding the neonatal environment, and reflecting on their service expectations. Based on father's/partner's preference, interviews will be undertaken either in a private room on the NU or virtually via MS Teams at a mutually convenient time. Interviews will be digitally recorded and are anticipated to last up to one hour. Data saturation is expected at around 12-15 fathers.
4. The parents will be asked to complete the PSS:NICU, GAD7 and PHQ9 questionnaires at 3 weekly intervals, finishing on the week of discharge, to monitor their MH through their NU stay.
5. Up to 4 groups of 5 mothers will be invited to participate in a focus group to assess their wellbeing, experience of the NU and their perspective on support for and from their partners. This will occur in a room in the NU at a time convenient to the mothers. Groups will be organised until data saturation is reached.
6. Telephone/online questionnaires will be completed by parents at 4-6 weeks post-discharge to assess family confidence and bonding after NU discharge.

Washout, Phase 2 Preparation: 4 months

1. The existing Neonatal DadPad app/booklet (which is currently used in several NHS Trusts to guide fathers through their NU journey) will be updated using phase-1 and systematic review study findings with guidance from the PAG, and a programme to enhance father participation within the FICare model will be developed.
2. Teaching sessions undertaken to educate and upskill all clinical NU staff on study aims, recruitment, phase-1 study findings and upcoming phase-2 study, highlighting the importance of fathers' role in the FICare (e.g., teaching parents how to safely give nasogastric feeds, nappy changes in a ventilated baby).

Phase 2 study. Enhanced Father involvement in FICare: 9 months. Once a family is recruited, the programme developed to enhance father involvement in FICare will be implemented to take place at the parents' pace. The NU experience and MH status of both parents will be assessed as in phase-1 study. At the end of phase-2 study, staff knowledge, experiences and opinions about fathers and FICare will be re-assessed and compared to the start of the study.

ELIGIBILITY:
Parents of preterm infants will be recruited to the study.

Inclusion criteria:

1. Parents of 22+0 to 32+6 weeks preterm infants.
2. Infant from day one to 7 days of age.
3. Infant should have two primary caregivers. Father's/Partner's participation in the study is a must and participation from both parents is ideal.
4. The parents should have conversational English.

Exclusion criteria:

1. Infant with life-limiting condition or no realistic chance of survival.
2. Infant is likely to be transferred to non-participating centre within 4 weeks of age.
3. Parents under the age of 16 years.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Babies born between 22+0 and 32+6 weeks who have two main caregivers
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Paternal mental health | From 1st week of baby's admission to discharge from the Neonatal Unit, up to 22 weeks
  Fathers' mental stress is assessed by semi-structured interviews.

SECONDARY OUTCOMES:
Fathers care giving ability | From 1st week of baby's admission to Neonatal Unit up to 6 weeks post discharge
  This will be assessed through semi-structured interview process.
Parental enagement | 6 weeks post baby discharge from Neonatal Unit
  This will be assessed by telephone interview at 6 weeks after baby's discharge fromneonatal unit.
Maternal mental health | From 1st week of baby's admission to Neonatal Unit up to 6 weeks post discharge
  Maternal stressor will be assessed by the PSS:NICU questionnaire
Paternal mental health | From 1st week of baby's admission to Neonatal Unit up to 6 weeks post discharge
  Parental stressor will be assessed by the PSS:NICU questionnaire.
Paternal anxiety | From 1st week of baby's admission to Neonatal Unit up to 6 weeks post discharge
  Paternal anxiety will be assessed by Generalised Anxiety Disorder Assessment-7
Paternal depression | From 1st week of baby's admission to Neonatal Unit up to 6 weeks post discharge
  Paternal depression will be assessed by the Personal Health Questionnaire-9

CONTACTS AND LOCATIONS:
Overall Officials: Narendra Aladangady, PhD, Study Director — Homerton Healthcare NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Neonatal Unit, Whipps Cross University Hospital, London
  - Neonatal Unit, Homerton University Hospital, London

IPD SHARING:
Plan to Share IPD: No
Anonymised data only collected

REFERENCES:
- [Derived] Rubinstein R, Gallagher K, Ho J, Bose J, Khashu M, Aladangady N. Investigating Father or Partner Involvement in Family Integrated Care in Neonatal Units: Protocol for a Prospective, Multicenter, Multiphase Study. JMIR Res Protoc. 2024 Mar 25;13:e53160. doi: 10.2196/53160. PMID 38526549